CLINICAL TRIAL: NCT05604521
Title: A Randomized, Double-blind, Placebo-controlled, Clinical Trial of a 3-dose, 28-day Regimen of PfSPZ Vaccine in Healthy, Adult Participants to Determine Safety, Tolerability and Efficacy Against Heterologous Plasmodium Falciparum Controlled Human Malaria Infection Conducted 3 or 12 Weeks After Immunization
Brief Title: A Phase 1 Trial of PfSPZ Vaccine in Healthy Adults to Determine Safety, Tolerability and Efficacy Against Heterologous CHMI
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The main reason for trial discontinuation was the inability to address the primary objectives of the study following an extended gap between the second and third doses.
Sponsor: Sanaria Inc. (Industry)
Collaborators: University of Maryland, Baltimore (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: USSPZV7; 1U44AI167783-01 (NIH)
Record Dates: First submitted 2022-10-28; First posted 2022-11-03 (Actual); Results first posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Malaria; Malaria,Falciparum
Keywords: Malaria; Plasmodium falciparum; Sporozoites; PfSPZ Vaccine
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1a: PfSPZ Vaccine (Active Comparator): 45 participants will receive 3 doses of 9.0x10^5 PfSPZ Vaccine on Days 1, 8, and 29 with a total dose of 2.7x10^6 PfSPZ Vaccine.
  Group 1a: Approximately half (22/23) of the volunteers will undergo CHMI 3 weeks after last immunization by exposure to 3.2x10^3 PfSPZ Challenge (7G8).
  Interventions: Biological: PfSPZ Vaccine; Biological: PfSPZ Challenge (7G8)
- Group 1b: PfSPZ Vaccine (Active Comparator): 45 participants will receive 3 doses of 9.0x10^5 PfSPZ Vaccine on Days 1, 8, and 29 with a total dose of 2.7x10^6 PfSPZ Vaccine.
  Group 1b: Approximately half (22/23) of the volunteers will undergo CHMI 12 weeks after last immunization by exposure to 3.2x10^3 PfSPZ Challenge (7G8).
  Interventions: Biological: PfSPZ Vaccine; Biological: PfSPZ Challenge (7G8)
- Group 2a: Normal Saline Controls (Placebo Comparator): 15 participants will receive 3 doses of normal saline on Days 1, 8, and 29.
  Group 2a: Approximately half (7/8) of the volunteers will undergo CHMI 3 weeks after last immunization by exposure to 3.2x10^3 PfSPZ Challenge (7G8).
  Interventions: Biological: PfSPZ Challenge (7G8); Other: Normal Saline
- Group 2b: Normal Saline Controls (Placebo Comparator): 15 participants will receive 3 doses of normal saline on Days 1, 8, and 29.
  Group 2b: Approximately half (7/8) of the volunteers will undergo CHMI 12 weeks after last immunization by exposure to 3.2x10^3 PfSPZ Challenge (7G8).
  Interventions: Biological: PfSPZ Challenge (7G8); Other: Normal Saline

INTERVENTIONS:
Biological: PfSPZ Vaccine — PfSPZ vaccine consists of radiation-attenuated, aseptic, purified Plasmodium falciparum (NF54) sporozoites (SPZ) cryopreserved in liquid nitrogen vapor phase (LNVP) at -150C to - 196C. PfSPZ Vaccine is composed of PfSPZ derived from the NF54 strain of Pf, which is thought to be from West Africa. PfSPZ Vaccine is diluted in phosphate buffered saline (PBS) with human serum albumin (HSA) to achieve the correct dosage and is administered by DVI.
  Arms: Group 1a: PfSPZ Vaccine; Group 1b: PfSPZ Vaccine
Biological: PfSPZ Challenge (7G8) — PfSPZ Challenge (7G8) is similar to PfSPZ Vaccine but has not been attenuated by radiation and is therefore infectious.PfSPZ Challenge (7G8) is composed of PfSPZ derived from the 7G8 clone of Pf, which is from Brazil.
Other: Normal Saline — 0.9% sodium chloride
  Other Names: Placebo
  Arms: Group 2a: Normal Saline Controls; Group 2b: Normal Saline Controls

SUMMARY:
USSPZV7 is a randomized, phase 1, double-blind, placebo-controlled trial of Sanaria® PfSPZ Vaccine administered on Days 1, 8 and 29 by direct venous inoculation (DVI) to assess safety, tolerability, immunogenicity, and vaccine efficacy (VE) against heterologous controlled human malaria infection (CHMI) with the 7G8 clone of Plasmodium falciparum (Pf) conducted at 3 or 12 weeks after the third immunization. The trial is designed to determine if individuals living in a non-malaria endemic area such as the United States (US) are protected against heterologous CHMI conducted at these time points.

DETAILED DESCRIPTION:
1. Randomized, phase 1, double-blind, placebo-controlled clinical trial enrolling healthy adult participants 18-50-years-old living in the US.
2. The trial is designed to measure safety, tolerability, immunogenicity and VE against heterologous controlled human malaria vaccine conducted at 3 or 12 weeks after vaccination.
3. Participants will be randomized to two study groups, vaccine and placebo, in a 3:1 ratio. Treatment assignment will be double blind; however, whether a given participant will be receiving CHMI at 3 or 12 weeks will not be blind.
4. Bias will be minimized by the randomized, double-blind design and by the inability to distinguish vaccine or placebo based on appearance, tolerability or other characteristics discernable by clinical staff or study participants.
5. The study will take approximately 6 to 8 months to complete, not including 2-3 months of recruitment. The period of follow-up for each immunized participant and placebo controls is through 8 weeks post-CHMI.
6. Study participation by individuals will last 4 to 6 months (not including screening) depending upon group assignment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults (male or non-pregnant female) 18 to 50 years of age.
* Able and willing to participate for the duration of the study.
* Able and willing to provide written informed consent and satisfactorily complete a test of understanding with a passing score >80%.
* Physical examination and laboratory results without clinically significant findings.
* Women of childbearing potential must agree to use effective means of birth control (e.g. oral or implanted contraceptives, IUD, female condom, diaphragm with spermicide, cervical cap, abstinence, use of a condom by the sexual partner or sterile sexual partner) during the entire study. Women with a history of surgical or chemical sterilization (e.g. tubal ligation, hysterectomy, other).
* Willing to refrain from blood donation for 3 years following CHMI.
* Agree not to travel to a malaria endemic region during the trial.

Exclusion Criteria:

* Unable to provide informed consent including inability to pass the test of understanding, which is written in English for the US-based study sites.
* Receipt of a malaria vaccine in a prior clinical trial.
* History of a splenectomy or sickle cell disease.
* History of a neurologic disorder (including non-febrile seizures or complex febrile seizures) or formal history of migraine headache.
* Current use of systemic immunosuppressant pharmacotherapy.
* Receipt of a live vaccine within 4 weeks of first immunization or of 3 or more non-live vaccines within 2 weeks of first immunization.
* Women who are breast-feeding, pregnant or planning to become pregnant during the study period.
* Known allergy to atovaquone-proguanil (Malarone®), artemether-lumefantrine (Coartem®), or any component of the investigational products.
* A history of malaria in the 2 years prior to screening.
* Participation in any study involving investigational vaccine or drug within 4 weeks prior to enrollment that in the estimation of the site PI might adversely affect the individual's safety or the quality of data to be collected.
* Evidence of increased cardiovascular disease risk; defined as >10% five-year risk by nonlaboratory method.
* Plan to participate in another investigational vaccine/drug research during the study.
* Plan for major surgery between enrollment until 28 days post-CHMI.
* Use or planned use of any drug with anti-malarial activity that would precede or coincide with malaria challenge or vaccination.
* Anticipated use of medications known to cause drug reactions with atovaquone-proguanil or artemether-lumefantrine such as cimetidine, metoclopramide, antacids, and kaolin.
* Positive HBsAg or positive HIV or HCV testing consistent with active infection.
* An abnormal electrocardiogram, defined as one showing pathologic Q waves and significant STT wave changes; left ventricular hypertrophy; any non-sinus rhythm including isolated premature ventricular contractions, but excluding isolated premature atrial contractions; right or left bundle branch block; or advanced (secondary or tertiary) A-V heart block; or other clinically significant abnormalities on the electrocardiogram as determined by the consulting cardiologist.
* Any clinically significant deviation from the normal range in biochemistry or hematology tests measured at screening and not resolving.
* Any medical, psychiatric, social, behavioral or occupational condition or situation (including active alcohol or drug abuse) that, in the judgment of the site PI, impairs the volunteer's ability to give informed consent, increases the risk to the participant of participation in the study, affects the ability of the participant to participate fully in the study, or might negatively impact the quality, consistency, integrity or interpretation of data derived from their participation in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy adults (male or non-pregnant female).
Enrollment: 31 (Actual)
Dates: Start 2022-12-06 (Actual); Primary Completion 2023-09-05 (Actual); Study Completion 2023-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten E Lyke, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore, Center for Vaccine Development and Global Health, Baltimore, Maryland, United States

REFERENCES:
- [Background] Mordmuller B, Sulyok Z, Sulyok M, Molnar Z, Lalremruata A, Calle CL, Bayon PG, Esen M, Gmeiner M, Held J, Heimann HL, Woldearegai TG, Ibanez J, Flugge J, Fendel R, Kreidenweiss A, Kc N, Murshedkar T, Chakravarty S, Riyahi P, Billingsley PF, Church LWP, Richie TL, Sim BKL, Hoffman SL, Kremsner PG. A PfSPZ vaccine immunization regimen equally protective against homologous and heterologous controlled human malaria infection. NPJ Vaccines. 2022 Aug 23;7(1):100. doi: 10.1038/s41541-022-00510-z. PMID 35999221
- [Background] Lyke KE, Singer A, Berry AA, Reyes S, Chakravarty S, James ER, Billingsley PF, Gunasekera A, Manoj A, Murshedkar T, Laurens MB, Church WP, Garver Baldwin LS, Sedegah M, Banania G, Ganeshan H, Guzman I, Reyes A, Wong M, Belmonte A, Ozemoya A, Belmonte M, Huang J, Villasante E, Sim BKL, Hoffman SL, Richie TL, Epstein JE; Warfighter II Study Team. Multidose Priming and Delayed Boosting Improve Plasmodium falciparum Sporozoite Vaccine Efficacy Against Heterologous P. falciparum Controlled Human Malaria Infection. Clin Infect Dis. 2021 Oct 5;73(7):e2424-e2435. doi: 10.1093/cid/ciaa1294. PMID 32920641
- [Derived] Berry AA, Richie TL, Church LWP, Laurens MB, Boyce C, Kc N, Joshi S, Koudjra AR, Butler L, Chen MC, Abebe Y, Murshedkar T, James ER, Billingsley PF, Sim BKL, Hoffman SL, Lyke KE. Safety, tolerability and immunogenicity of a condensed, multi-dose prime regimen of PfSPZ Vaccine for the prevention of Plasmodium falciparum malaria infection. Malar J. 2025 Mar 17;24(1):88. doi: 10.1186/s12936-025-05299-5. PMID 40098097

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Altogether, 72 persons were screened, 31 received immunizations, 15 were screen failures, 4 were eligible but yet not enrolled, and 22 were still being evaluated when the study was terminated.
Groups:
- Group 1: PfSPZ Vaccine: N=24; received at least 1 dose of vaccine.
- Group 2: Normal Saline Placebo: N=7; received normal saline placebo
Period: Overall Study
Arm/Group | Group 1: PfSPZ Vaccine | Group 2: Normal Saline Placebo
Started | 24 | 7
Completed | 0 | 0
Not Completed | 24 | 7
Not completed — Trial terminated early due to an extended gap between the 2nd and 3rd doses (3rd dose not given). | 23 | 7
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: PfSPZ Vaccine | Group 2: Normal Saline Placebo | Total
Number analyzed (Participants) | 24 | 7 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 7 | 31
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 3 | 13
  Male | 14 | 4 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 18 | 6 | 24
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 7 | 31

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: The differences in proportions of vaccinees compared to controls experiencing related moderate, severe, or serious solicited and unsolicited adverse events and laboratory abnormalities after vaccination.
Time Frame: Day of immunization to 28 days post immunization
Population: 24 participants received a 1st dose and 23 participants received a 2nd dose of vaccine, and 7 participants received 2 doses of placebo. Due to early study termination, we measured outcome variables for which data were available: proportion of participants experiencing local solicited AEs, systemic solicited AEs and related unsolicited AEs.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: PfSPZ Vaccine | Group 2: Normal Saline Placebo
Number analyzed (Participants) | 24 | 7
Participants | 17 | 7
Statistical Analysis 1: Comparison: Group 1: PfSPZ Vaccine vs Group 2: Normal Saline Placebo; Null hypothesis: There is no statistically significant difference between the vaccine and control groups in the proportion of participants experiencing any local solicited AEs after any vaccination; Test type: Superiority; p = 0.3944, Fisher Exact
Statistical Analysis 2: Comparison: Group 1: PfSPZ Vaccine vs Group 2: Normal Saline Placebo; Null hypothesis: There is no statistically significant difference between the vaccine and control groups in the proportion of participants experiencing any systemic solicited AEs after any vaccination; Test type: Superiority; p = 0.3717, Fisher Exact
Statistical Analysis 3: Comparison: Group 1: PfSPZ Vaccine vs Group 2: Normal Saline Placebo; Null hypothesis: There is no statistically significant difference between the vaccine and control groups in the proportion of participants experiencing any related unsolicited AEs after any vaccination; Test type: Superiority; p = 1.0, Fisher Exact

ADVERSE EVENTS:
Time Frame: Solicited local adverse events (AEs) were collected for two days after each immunization. Solicited systemic AEs were collected for 7 days after each immunization. Unsolicited AEs were collected from the first immunization to 28 days after the second immunization (since the study was terminated early). SAEs were to be recorded through the entire duration of the trial.
Description: Solicited local AEs: pain & pruritus (by questioning participant), tenderness & induration (by palpation) & erythema, bruising & swelling (by visual inspection, swelling by viewing site laterally for swelling of skin). Solicited systemic AEs: fever (oral temp > 100.4 F), subjective fever, chills, headache, fatigue, malaise, myalgia, arthralgia, rigors, systemic allergic type reactions (rash, urticaria, pruritus, edema). Unsolicited AEs: open-ended question (e.g.do you have any other symptoms?).
Arm/Group | Group 1: PfSPZ Vaccine | Group 2: Normal Saline Placebo
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/7
Other Adverse Events (participants affected / at risk) | 17/24 | 7/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: PfSPZ Vaccine (N=24) | Group 2: Normal Saline Placebo (N=7)
Allergic reaction - hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) — Unsolicited AE; related.
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) — Unsolicited AE; related.
Bruising (General disorders) | 7 (9) | 5 (8) — Solicited local AE
Erythema (General disorders) | 5 (6) | 4 (4) — Solicited local AE
Pain (General disorders) | 3 (3) | 2 (2) — Solicited local AE
Swelling (General disorders) | 1 (1) | 1 (1) — Solicited local AE
Tenderness (General disorders) | 1 (1) | 0 (0) — Solicited local AE
Fatigue (General disorders) | 8 (8) | 4 (4) — Solicited systemic AE
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0) — Solicited systemic AE
Chills (General disorders) | 4 (4) | 1 (1) — Solicited systemic AE
Subjective fever (General disorders) | 6 (6) | 2 (2) — Solicited systemic AE
Headache (Nervous system disorders) | 9 (12) | 3 (3) — Solicited systemic AE
Malaise (General disorders) | 7 (9) | 3 (3) — Solicited systemic AE
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (11) | 4 (5) — Solicited systemic AE
Rigors (General disorders) | 5 (5) | 1 (1) — Solicited systemic AE
Systemic allergic type reaction - dermatographia (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) — Solicited systemic AE
Systemic allergic type reaction - feet pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Solicited systemic AE
Fever (General disorders) | 1 (1) | 1 (1) — Solicited systemic AE

LIMITATIONS AND CAVEATS:
The trial was terminated early. The main reason for trial discontinuation was the inability to address the primary objectives of the study following an extended gap between the second and third doses. Thus, vaccination was not completed and efficacy measurement was not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
(1) The principal investigator and associated institution are restricted from using the results of the study for commercial purposes; (2) the principal investigator is obligated to provide the Sponsor an opportunity to review planned disseminations of the data for "confidential information" that if present must be removed on Sponsor's request; (3) it is stipulated that communications such as publications and presentations should be "joint."

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-21): https://cdn.clinicaltrials.gov/large-docs/21/NCT05604521/Prot_SAP_000.pdf